CLINICAL TRIAL: NCT00287690
Title: The Effect of Genistein (Supro®) on Coronary Artery Diameter and Blood Flow in Men and Women With Coronary Heart Disease
Brief Title: Isoflavones and the Coronary Circulation in Men and Women With Coronary Artery Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 98-170
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2006-02

CONDITIONS: Coronary Artery Disease
Keywords: arteries; blood flow; coronary artery disease; diet
MeSH Terms: conditions — Coronary Artery Disease | interventions — Genistein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Genistein (Experimental): Supro drink once daily for 3 days
  Interventions: Drug: Genistein
- Placebo (Placebo Comparator): Drink identical to Supro but containing no genistein, once daily for 3 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Genistein — Drink taken once daily
  Other Names: Supro
  Arms: Genistein
Drug: Placebo — Drink taken once daily
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the effect of genistein administration on coronary arteries in humans. We will measure the size of a coronary artery and the speed and amount of blood flow in response after subjects have ingested Supro® drinks (a soy protein drink containing genistein).

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-75 years
* Patients requiring diagnostic coronary angiography
* Presence of coronary artery disease on angiogram but with at least one non-obstructed (lesions <70% narrowed compared with the adjacent normal part of the vessel) atheromatous vessel (confirmed at diagnostic cardiac catheterisation)
* Female patients must be postmenopausal (FSH>40 IU/L)
* Willing to give informed, written consent

Exclusion Criteria:

* Age <30 or >75 years
* Allergy to radiographic contrast media
* Sino-atrial disease or significant bradycardia
* Concomitant medication with persantin (dipyridamole) or theophyllines
* Asthma
* Hypertension
* Left ventricular hypertrophy or dysfunction (clinical/ECG/echo/CXR)
* Female patients with FSH<40 IU/L (postmenopausal)
* Female patients currently taking hormone therapy, or who have taken hormone therapy in previous 6 months
* Unwilling to give written informed consent
* Participation in another study within previous 60 days

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 1999-10; Primary Completion 2003-08-18 (Actual); Study Completion 2003-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Collins, MD, FRCP, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton & Harefield NHS Trust, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Genistein: Supro drink once daily for 3 days prior to coronary angiography
  Genistein: Drink taken once daily
- Placebo: Drink identical to Supro but containing no genistein, once daily for 3 days prior to coronary angiography.
  Placebo: Drink taken once daily
Period: Overall Study
Arm/Group | Genistein | Placebo
Started | 33 | 38
Completed | 13 | 12
Not Completed | 20 | 26
Not completed — Protocol Violation | 20 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genistein | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 9 | 22
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 13 | 9 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Coronary Artery Diameter
Description: Coronary angiograms were acquired digitally using a real-time digital image acquisition system (Siemens AG, Berlin and Munich, Germany) and analysed off-line using quantitative coronary angiography (MEDIS, Leiden, The Netherlands). Basal luminal diameter of the entire coronary artery (mean luminal diameter) was measured for all subjects. Mean luminal diameter and luminal diameter approximately 4 mm distal to the tip of the Doppler wire were measured. The latter measurements were used to quantify volume flow as described previously. Data below are mean coronary artery diameter response following infusion of acetylcholine (ACh 10-5 M).
Time Frame: Day 3-4 after Supro/placebo started.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Genistein | Placebo
Number analyzed (Participants) | 13 | 12
mm | 3.1 (0.4) | 2.7 (0.4)

2. Primary Outcome: Coronary Blood Flow
Description: Measurement of diameter 4mm distal to the Doppler wire tip (measured using quantitative coronary angiography) and blood flow velocity, measured using intracoronary Doppler), were made at baseline and at peak velocity change. A quantitative estimate of coronary blood flow was calculated from the Doppler flow velocity and quantitative angiographic data using the following equation: Q = 3.14(D2/4)(APV/2)(0.6) where Q is flow (ml/min), D is vessel diameter (mm) and APV is average peak velocity (cm/s). Data below are measurements taken at peak blood flow response following an infusion of acetylcholine (10-5M).
Time Frame: Day 3-4 after Supro/placebo started.
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Genistein | Placebo
Number analyzed (Participants) | 13 | 12
ml/min | 77 (34) | 68 (32)

3. Secondary Outcome: Serum Genistein Concentrations
Description: Measured from serum using liquid-chromatographic tandem mass spectrometric bioanalytical assays (HFL Ltd, Fordham, Cambridgeshire, UK).
Time Frame: Day 3 after Supro/placebo started.
Measure: Median (95% Confidence Interval); unit: ng/ml
Arm/Group | Genistein | Placebo
Number analyzed (Participants) | 13 | 12
ng/ml | 340 [247 to 515] | 3.9 [1.7 to 5.8]

ADVERSE EVENTS:
Time Frame: From enrollment to study end, approximately 1 week.
Arm/Group | Genistein | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes